CLINICAL TRIAL: NCT01536548
Title: Indicating Direction and Angle for Button-hole Cannulating of AV-fistula in Hemodialysis Patients - a Randomized Controlled Study
Brief Title: Indicating Direction and Angle for Cannulating of AV-fistula in Hemodialysis Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian University of Science and Technology (Other)
Collaborators: St. Olavs Hospital (Other); Haukeland University Hospital (Other); Vestre Viken Hospital Trust (Other); Sykehuset Innlandet HF (Other); Kristiansund Hospital (Other); Bodø sykehus (Unknown); University Hospital, Akershus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2011/2544
Record Dates: First submitted 2012-02-16; First posted 2012-02-22 (Estimated); Last update posted 2020-10-05 (Actual); Status verified 2020-09

CONDITIONS: Chronic Kidney Disease; Kidney Failure
Keywords: hemodialysis; cannulation; AV-fistula; buttonhole technique
MeSH Terms: conditions — Renal Insufficiency, Chronic; Renal Insufficiency; Arteriovenous Fistula

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Skin drawing (Experimental)
  Interventions: Procedure: Skin drawing
- No skin drawing (Active Comparator)
  Interventions: Procedure: No skin drawing

INTERVENTIONS:
Procedure: Skin drawing — Mark direction and angle for cannulation with a pencil on the skin
  Arms: Skin drawing
Procedure: No skin drawing — Standard practice; i.e. no marks on skin to help find correct direction and angle for introducing needles
  Arms: No skin drawing

SUMMARY:
Arteriovenous fistula is the preferred access for hemodialysis, and cannulation using a "button-hole" technique is increasingly recommended. By using the same two sites for cannulation there are reports of less risk of complications and less pain for the patient. However, button-hole cannulation can be difficult for the dialysis nurse, and failing cannulations can damage the AV fistula and increase patient discomfort. The investigators therefore will test whether a simple marking on the skin of the direction and angle of cannulation used in each specific patient could improve the probability of a successful and painfree cannulation.

ELIGIBILITY:
Inclusion Criteria:

* chronic kidney disease
* hemodialysis
* arteriovenous fistula
* established buttonhole technique
* informed consent signed

Exclusion Criteria:

* child
* minor
* not speaking Norwegian
* not willing to sign informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2012-03; Primary Completion 2012-04 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Percentage of successful cannulations | 8 weeks
  A successful cannulation is defined as being able to insert a blunt needle in both canals at the first attempt.

SECONDARY OUTCOMES:
Difficulty of cannulation | 8 weeks
  Nurse and patients describe on a Verbal Rating Scale (1-6) how difficult the cannulation was experienced. All dialysis sessions are scored.
Fear of cannulation | 8 weeks
  Patients describe on a Verbal Rating Scale (0-10) how strongly they fear the cannulation. Assessed once a week.
Pain at cannulation | 8 weeks
  Patients describe on a VAS scale (0-10) how painful the cannulation was experienced. Assessed once a week.

CONTACTS AND LOCATIONS:
Overall Officials: Stein Hallan, PhD MD, Study Director — Norwegian University of Science and Technology
Locations (8):
- Norway (8):
  - Haukeland Universitetssykehus, Bergen
  - Bodø Sykehus, Bodø
  - Vestre Viken Sykehus, Drammen
  - Kristiansund Sykehus, Kristiansund
  - Sykehuset Innlandet, Lillehammer
  - St Olavs Hospital, Orkanger
  - Akershus Universitetssykehus, Oslo
  - St Olavs Hospital, Trondheim

REFERENCES:
- [Background] Rønning MI, Benshop P , Hallan S. Direction and angle-assisted cannulation of AV-fistula in hemodialysis patients - a rancomized controlled study. 2016; Oral presentation for the Vascular Access Society of America, Chicago 2016, abstract 1.1.4.8
- [Derived] Ronning MI, Benschop WP, Ovrehus MA, Hultstrom M, Hallan SI. Direction- and Angle-Assisted Buttonhole Cannulation of Arteriovenous Fistula in Hemodialysis Patients: A Multicenter Randomized Controlled Trial. Kidney Med. 2021 Dec 1;4(2):100393. doi: 10.1016/j.xkme.2021.10.006. eCollection 2022 Feb. PMID 35243305